CLINICAL TRIAL: NCT04464551
Title: A Single-center, Open-label, Single-dose Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C]D-0316 After a Single Oral 75mg/50µCi Dose in Healthy Chinese Male Subjects
Brief Title: The Absorption, Metabolism and Excretion of [14C]D-0316 in Human
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBIO-105
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Advanced or Metastatic Non-small Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]D-0316 (Experimental): To investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose (75mg, 50µCi) of [14C]D-0316 to healthy Chinese male subjects
  Interventions: Drug: [14C]D-0316 suspension

INTERVENTIONS:
Drug: [14C]D-0316 suspension — Before administration, the drug preparation was placed at room temperature, and 40ml drinking water was added into each bottle to prepare suspension for the subjects to take. 40ml pure water was injected again. After washing the container, the subjects took orally. Repeat the previous step, and then used 160ml purified water. After the administration container was moistened for several times, the subjects took all the moistening lotion. Pay attention not to splash the liquid during mixing outside the bottle

SUMMARY:
This is a single-center, open-label, single-dose phase I study to investigate the absorption, metabolism and excretion of [14C] D-0316 in healthy Chinese male subjects. The study will be conducted into two steps：Firstly, 2 subjects are enrolled in to participate in the pilot study to grope for the completion date of plasma, urine and feces sampling on the 3rd day post-dose and onwards. Then, the collection time of blood and excreta samples (urine and feces) from the subsequent 2-4 subjects will be adjusted according to the pilot study

DETAILED DESCRIPTION:
Subjects who had signed informed consent and meet inclusion criteria and no exclusion criteria are admitted to Phase I Clinical Unit two days prior to dosing (D-2). On the morning of Day 1 before dosing, subjects will be transferred to nuclear medical ward. And after an overnight fast of at least 10 h, subjects will receive a single oral dose of 75 mg (50 μCi) of [14C]D-0316 as an oral suspension. Then, after two days of the dosing, subjects will be transferred back to Phase I Clinical Unit ward and confined to this unit until blood or excreta sampling and safety monitoring at the designated time points or intervals are complete

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers between the ages of 18 to 50 years old；
* Body weight >=50 kg, Body mass index (body weight(kg)/hight2(m2)) between 19 and 26 kg/m2；
* Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant;
* Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 1 year after discontinuing treatment with the investigational product. Highly effective methods of birth control include using condom, contraceptive sponge, contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptive pill, hypodermic implants or others；
* Must understand, and voluntarily sign the informed consent, comply with the requirements of the study.

Exclusion Criteria:

* History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder;
* Positive test for HBsAg, HBeAg, anti-HCV, anti-HIV or syphilis antibody;
* History of syncope / needle syncope and intolerable intravenous indwelling needle;
* History of clinically significant disease or infection within 1 month before entering the study;
* Abnormality in blood pressure, including hypertensive BP (SBP>=140 mmHg, or DBP >=90 mmHg), or hypotensive BP(SBP<90 mmHg, or DBP <=55 mmHg), Pulse rate<55 bpm or >100 bpm;
* Long-QT syndrome or family history of it, or QTcB interval > 450 ms; intraventricular blocks or left/right bundle branch block or QRS>120ms; frequent ventricular ectopic beats (any 10s ECG ventricular premature beat >= 1 in screening period); or abnormal resting heart rate (> 100 bpm);
* Received any drug within 14 days before taking the investigational drug, including any prescription drug, OTC drug, herbal drug or health care products, except for vitamins and paracetamol；
* History of or current swallowing disorder, active gastrointestinal diseases, or other diseases that significantly affect absorption, distribution, metabolism and excretion of drugs;
* Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
* Hemorrhoids or perianal disease with regular/perianal bleeding;
* Allergies, have allergies to two or more drugs or foods; or have known allergies to the components of the drug;
* Participated in other clinical trials within 3 months before screening;
* The subjects participated in the clinical trial of radioactive labeling within one year before taking the medicine;
* Significant radiation exposure within one year prior to drug administration (more than one exposure from chest X-ray, CT scan, or barium meal examination and radiation-related occupations);

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Radioactivity concentration of each plasma sample | Day 1-Day85
  Use liquid scintillation counter or accelerator mass spectrometry to evaluate radioactivity concentration of each plasma（DPM/ml) sample
Radioactivity concentration of each urine samples | Day-1-Day85
  Use liquid scintillation counter or accelerator mass spectrometry to evaluate radioactivity concentration of each urine（DPM/ml) sample
Radioactivity concentration of each feces sample | Day-1-Day85
  Use liquid scintillation counter or accelerator mass spectrometry to evaluate radioactivity concentration of each feces（DPM/ml) sample
Total recovery of radioactivity in urine and feces | Day-1-Day85
  Calculate the total radioactivity in urine and feces based on the radioactivity concentration of each sample
Identification of metabolites in plasma, urine and fecal samples | Day-1-Day85
  LC-MS/MS was used to identify the main metabolites in plasma, urine and feces, and finally to provide the main biotransformation pathway of CM082 in human body

SECONDARY OUTCOMES:
Pharmacokinetic parameters of unlabeled D-0316 and metabolite D-0865 | Day-1-Day85
  To determine the plasma concentrations of D-0316 with validated LC-MS/MS method for obtaining its pharmacokinetics parameters
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Day-14-Day85
  According to CTCAE v4.03, the number and frequency of adverse events after a single dose of test drug were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Ph D, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine; Wei Liu, M.A, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine
Locations (1):
- Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine, Nanjing, Jiangsu, China